CLINICAL TRIAL: NCT02086500
Title: Study of Tranexamic Acid During Air and Ground Medical Prehospital Transport Trial For Trauma Patients At Risk Of Hemorrhage (STAAMP Trial); Phase III Multicenter, Prospective, Randomized, Double Blind, Interventional Trial
Brief Title: Study of Tranexamic Acid During Air and Ground Medical Prehospital Transport Trial (STAAMP Trial)
Acronym: STAAMP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jason Sperry (Other)
Collaborators: University of Arizona (Other); The University of Texas at San Antonio (Other); University of Utah (Other)
Responsible Party: Sponsor-Investigator, Jason Sperry, MD, MPH, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: W81XWH1320080 IND 121102
Record Dates: First submitted 2014-03-06; First posted 2014-03-13 (Estimated); Results first posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Traumatic Hemorrhage
Keywords: Tranexamic acid; randomized; hemorrhage; blinded
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prehospital Tranexamic Acid (Experimental): 1 gram of Tranexamic Acid will be given during emergency medical transport
  Interventions: Drug: Tranexamic Acid
- Control (Placebo Comparator): Identical volume of saline during emergency medical transport
  Interventions: Other: Saline control

INTERVENTIONS:
Drug: Tranexamic Acid — 1 gram of prehospital Tranexamic Acid
  Arms: Prehospital Tranexamic Acid
Other: Saline control — Saline Control
  Arms: Control

SUMMARY:
The purpose of this study is to determine if 1 gram of prehospital tranexamic acid given during emergency medical transport to a level 1 trauma center in patients at risk of hemorrhage is associated with lower 30 day mortality.

DETAILED DESCRIPTION:
Background: Traumatically injured patients continue to be plagued with uncontrolled hemorrhage resulting in significant morbidity and early mortality. A primary driving force for this unbridled hemorrhage is known to be the early coagulopathy which complicates severe injury. Trauma induced coagulopathy has been postulated to be an equilibrium imbalance between pro and anticoagulant factors, platelets, endothelium and fibrinolysis soon after injury. Recent evidence demonstrates that the early use of the antifibrinolytic agent tranexamic acid (TXA) after trauma center arrival results in improved survival in patients at risk for bleeding. Bringing this proven treatment to the prehospital arena and intervening earlier in those patients who would otherwise not be candidates for treatment has the real potential to further reduce or prevent the vicious hemorrhagic cascade, improve clinical outcomes and provide insight into the underlying mechanisms responsible for and which maximize its benefit.

Objective/Hypothesis: The primary hypothesis will be that prehospital infusion of tranexamic acid in patients at risk for bleeding will reduce the incidence of 30 day mortality. The secondary hypotheses include that prehospital tranexamic acid will reduce the incidence of hyperfibrinolysis, acute lung injury, multiple organ failure, nosocomial infection, mortality, early seizures, pulmonary embolism and early resuscitation needs, reduce or prevent the early coagulopathy as demonstrated by improving presenting INR and rapid thromboelastography parameters, reduce the early inflammatory response, plasmin levels, leukocyte, platelet and complement activation, and determine the optimal dosing of tranexamic acid post-injury.

ELIGIBILITY:
Inclusion Criteria:

1. Blunt or penetrating injured patients at risk of bleeding being transported via air or ground medical services from the scene of injury or from referring hospital to a definitive trauma center that is participating in the trial AND
2. Within 2 hours of time of injury AND
3. Hypotension (Systolic Blood Pressure (SBP) < 90mmHg)

   * At scene of injury or during air or ground medical transport
   * Documented at referring hospital prior to air or ground medical transport arrival

   OR
4. Tachycardia (heart rate >110 beats per minute)

   * At scene of injury or during air or ground medical transport
   * Documented at referring hospital prior to air or ground medical transport arrival

Exclusion Criteria:

1. Age > 90 or < 18 years of age
2. Inability to obtain intravenous access or intraosseous
3. Documented (radiographic evidence) cervical cord injury with motor deficit
4. Known prisoner
5. Known pregnancy
6. Traumatic arrest with > 5 minutes CPR without return of vital signs
7. Penetrating cranial injury
8. Traumatic brain injury with brain matter exposed
9. Isolated drowning or hanging victims
10. Wearing an opt out bracelet.
11. Isolated fall from standing
12. Patient or Family Objection at scene

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 903 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Lorence JM, Donohue JK, Iyanna N, Guyette FX, Gimbel E, Brown JB, Daley BJ, Eastridge BJ, Miller RS, Nirula R, Harbrecht BG, Claridge JA, Phelan HA, Vercruysse G, O'Keeffe T, Joseph B, Neal MD, Sperry JL. Characterization of adverse events in injured patients at risk of hemorrhagic shock: a secondary analysis of three harmonized prehospital randomized clinical trials. Trauma Surg Acute Care Open. 2024 Jun 25;9(1):e001465. doi: 10.1136/tsaco-2024-001465. eCollection 2024. PMID 38933603
- [Derived] Gruen DS, Brown JB, Guyette FX, Johansson PI, Stensballe J, Li SR, Leeper CM, Eastridge BJ, Nirula R, Vercruysse GA, O'Keeffe T, Joseph B, Neal MD, Sperry JL. Prehospital tranexamic acid is associated with a dose-dependent decrease in syndecan-1 after trauma: A secondary analysis of a prospective randomized trial. J Trauma Acute Care Surg. 2023 Nov 1;95(5):642-648. doi: 10.1097/TA.0000000000003955. Epub 2023 May 1. PMID 37125811
- [Derived] Guyette FX, Brown JB, Zenati MS, Early-Young BJ, Adams PW, Eastridge BJ, Nirula R, Vercruysse GA, O'Keeffe T, Joseph B, Alarcon LH, Callaway CW, Zuckerbraun BS, Neal MD, Forsythe RM, Rosengart MR, Billiar TR, Yealy DM, Peitzman AB, Sperry JL; STAAMP Study Group. Tranexamic Acid During Prehospital Transport in Patients at Risk for Hemorrhage After Injury: A Double-blind, Placebo-Controlled, Randomized Clinical Trial. JAMA Surg. 2020 Oct 5;156(1):11-20. doi: 10.1001/jamasurg.2020.4350. Online ahead of print. PMID 33016996

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prehospital Tranexamic Acid | Control
Started | 447 | 456
Completed | 447 | 456
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: of the 927 patients enrolled in the prehospital environment, 903 were able to be analyzed
Groups:
- Total: Total of all reporting groups
Arm/Group | Prehospital Tranexamic Acid | Control | Total
Number analyzed (Participants) | 447 | 456 | 903
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 39 [26 to 53] | 39 [26 to 56] | 39 [26 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 115 | 235
  Male | 327 | 341 | 668
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 2 | 3 | 5
  Black or African American | 49 | 40 | 89
  White | 353 | 361 | 714
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 41 | 49 | 90

OUTCOME MEASURES:

1. Primary Outcome: 30 Day Mortality
Description: Because not all patients had available data regarding 30-day mortality (patients were discharged and there 30-day outcome was unable to be determined) there may be differences between the 30Day mortality relative to the other outcomes. There were 5 and 4 patients from each arm that did not have 30-day outcome and thus are different.
Time Frame: 30 Day
Population: Because not all patients had available data regarding 30-day mortality (patients were discharged and there 30-day outcome was unable to be determined) there may be differences between the 30Day mortality relative to the other outcomes. There were 5 and 4 patients from each arm that did not have 30-day outcome and thus are different.
Measure: Count of Participants; unit: Participants
Arm/Group | Prehospital Tranexamic Acid | Control
Number analyzed (Participants) | 442 | 452
Participants | 36 | 45

2. Secondary Outcome: 24 Hour Mortality
Time Frame: 24 Hours
Measure: Count of Participants; unit: Participants
Arm/Group | Prehospital Tranexamic Acid | Control
Number analyzed (Participants) | 447 | 453
Participants | 16 | 17

3. Secondary Outcome: Acute Lung Injury
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Prehospital Tranexamic Acid | Control
Number analyzed (Participants) | 447 | 453
Participants | 42 | 39

4. Secondary Outcome: Multiple Organ Failure
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Prehospital Tranexamic Acid | Control
Number analyzed (Participants) | 447 | 453
Participants | 33 | 39

5. Secondary Outcome: Nosocomial Infection
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Prehospital Tranexamic Acid | Control
Number analyzed (Participants) | 447 | 453
Participants | 88 | 66

6. Secondary Outcome: 24 Hour Total Blood Transfusion
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: units of blood transfusion
Arm/Group | Prehospital Tranexamic Acid | Control
Number analyzed (Participants) | 447 | 453
units of blood transfusion | 0 [0 to 2] | 0 [0 to 2]

7. Secondary Outcome: Hyperfinbrinolysis
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Prehospital Tranexamic Acid | Control
Number analyzed (Participants) | 447 | 453
Participants | 145 | 144

ADVERSE EVENTS:
Time Frame: Hospital Admission to 30 days
Arm/Group | Prehospital Tranexamic Acid | Control
All-Cause Mortality (participants affected / at risk) | 36/447 | 45/456
Serious Adverse Events (participants affected / at risk) | 4/447 | 7/456
Other Adverse Events (participants affected / at risk) | 4/447 | 14/456
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prehospital Tranexamic Acid (N=447) | Control (N=456)
Stroke (Nervous system disorders) | 1 (1) | 2 (2) — Stroke
MI (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary Embolus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Arterial Thromboembolic event NOS (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prehospital Tranexamic Acid (N=447) | Control (N=456)
ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pnuemonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 2 (2)
Stroke (Nervous system disorders) | 0 (0) | 2 (2)
Venous Thromboembolic Event NOS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT02086500/Prot_SAP_000.pdf